CLINICAL TRIAL: NCT02263807
Title: RCT Study:Knee Function in Patients With Two or More Episodes of Patella Dislocations
Brief Title: Knee Function in Patients With Two or More Episodes of Patella Dislocations
Acronym: MPFL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asbjorn Aroen (Other)
Responsible Party: Sponsor-Investigator, Asbjorn Aroen, Professor, Orthopaedic Surgeon, University Hospital, Akershus
Organization: University Hospital, Akershus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009/2148
Record Dates: First submitted 2011-12-22; First posted 2014-10-13 (Estimated); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Joint Instability
Keywords: Patella luxation
MeSH Terms: conditions — Joint Instability | interventions — Arthroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MPFL group (Experimental): Arthroscopy and MPFL reconstruction
  Interventions: Procedure: MPFL Group; Procedure: Control
- Control (Active Comparator): Arhroscopy and rehabilitation
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: MPFL Group — MPFL reconstruction or standard treatment followed by physiotherapy
  Other Names: MPFL surgery
  Arms: MPFL group
Procedure: Control — Arthroscopy followed by active rehabilitation
  Other Names: Arthroscopy

SUMMARY:
Patients aged 12 - 30 years, with recurrent patella dislocations, are consecutively included into a randomized prospective study. This study comparess the outcome of two forms of treatment for recurrent patella dislocation. One group is offered reconstruction of the medial patellofemoral ligament (MPFL), the second group is offered a standardized training program.

DETAILED DESCRIPTION:
Introduction:

Patella dislocation is a serious knee injury whose peak incidence occurs in patients aged 10-17 years and is associated with a high rate of re-dislocation. Knee injuries frequently cause long-term disability and reduced physical activity among adolescents and young persons. Surgery in this patient group requires a low tolerance for complications, meaning that physical therapy might offer more successful outcomes in many knee injury cases. The proposed project studies a particular patient cohort subjected to recurrent dislocation of the patella.

Aim:

The principal objective of this clinical, randomized controlled trial is to evaluate and compare knee function and symptoms in patients with recurrent patella dislocation randomized into treatment with surgical reconstruction of the medial patellofemoral ligament (MPFL) with those of patients in a standardized physiotherapy program designed to stabilize the patella and improve patient function.

Materials and methods:

Patients aged 12-30 years who have experienced two or more patella dislocations are randomized into groups receiving either MPFL reconstruction or physical therapy only. Follow-ups at 3, 6, 12, and 36 months involve functional tests, validated knee scores, arthroscopic examination, and cartilage-specific MRI protocols for the knee.

ELIGIBILITY:
Inclusion Criteria:

* More than one luxation
* Norwegian citizens
* Unilateral problems
* Age range 12-30 years

Exclusion Criteria:

-Generalized degenerative changes

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Reoperation | 2011-2022
  Numbers of reoperation in the two treatment groups

SECONDARY OUTCOMES:
Patella reluxation | 2011-2022
  Number of reluxation of patella in the two treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn Årøen, MD,PhD, Study Chair — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lørenskog, Norway

REFERENCES:
- [Result] Straume-Naesheim TM, Randsborg PH, Mikaelsen JR, Sivertsen EA, Devitt B, Granan LP, Aroen A. Recurrent lateral patella dislocation affects knee function as much as ACL deficiency - however patients wait five times longer for treatment. BMC Musculoskelet Disord. 2019 Jul 8;20(1):318. doi: 10.1186/s12891-019-2689-7. PMID 31286929
- [Result] Straume-Naesheim TM, Randsborg PH, Mikaelsen JR, Aroen A. Medial patellofemoral ligament reconstruction is superior to active rehabilitation in protecting against further patella dislocations. Knee Surg Sports Traumatol Arthrosc. 2022 Oct;30(10):3428-3437. doi: 10.1007/s00167-022-06934-3. Epub 2022 Mar 28. PMID 35347375
- [Derived] Straume-Naesheim TM, Randsborg PH, Nilsgard TL, Aroen A. Medial Patellofemoral Ligament Reconstruction vs Nonoperative Treatment for Recurrent Lateral Patellar Dislocation: Three-Year Results From a Randomized Controlled Trial. Am J Sports Med. 2026 Feb 8:3635465261416931. doi: 10.1177/03635465261416931. Online ahead of print. PMID 41655186
- [Derived] Nilsgard TL, Oiestad BE, Randsborg PH, Aroen A, Straume-Naesheim TM. Association between single leg hop tests and patient reported outcome measures and patellar instability in patients with recurrent patellar dislocations. BMJ Open Sport Exerc Med. 2023 Dec 30;9(4):e001760. doi: 10.1136/bmjsem-2023-001760. eCollection 2023. PMID 38170085